CLINICAL TRIAL: NCT05349747
Title: Outcome of Treatment of Uveitis With Biologic Drugs in Resistant Cases Vogt-koyanagi-Harada Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Safwat Abdelhady Hafez, Assistant lecturer, Assiut University
Other Study IDs: Uveitis
Record Dates: First submitted 2022-04-11; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Biological Products

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Biological: Biologic drugs — Assess the results of treatment with biologic drugs

SUMMARY:
* Reviewing the characteristics of patients with uveitis caused by Vogt-Koyanagi-Harada Syndrome treated at Assiut University Hospital at the Department of Ophthalmology and Department of Rheumatology, Physical Medicine, and Rehabilitation including the ocular features in terms of uveitis location, type and complications and systemic features of those subjects who showed an inadequate response to conventional immunomodulatory drugs.
* Assess the results of treatment with biologic drugs, including rates of failure and adverse events. This will help uveitis specialists to reach a conclusion about the best treatment protocols for Uveitis in Vogt-Koyanagi-Harada Syndrome in our population in terms of safety, efficacy, and cost-effectiveness.

DETAILED DESCRIPTION:
Uvea (Latin for grape) is the middle vascular coat of the eyeball. Strictly speaking, uveitis is defined as inflammation of the uvea, but often the inflammatory process involves adjacent intraocular structures e.g. the anterior chamber, the vitreous humor, or the retina. Inflammation in the uvea can be due to infections, masquerades such as B-cell lymphoma, or immune-mediated diseases.

Vogt-Koyanagi-Harada syndrome is a systemic autoimmune disease characterized by bilateral, chronic, diffuse granulomatous panuveitis in addition to neurological, auditory, and integumentary manifestations. These manifestations are variable and race dependent.

This inflammatory syndrome is probably the result of an autoimmune mechanism, influenced by genetic factors, and appears to be directed against melanocytes. On histopathologic examination, typical cases show non-necrotizing diffuse granulomatous panuveitis with initial sparing and late involvement of the choriocapillaris and formation of Dalen-Fuchs' nodules. Fluorescein angiography, lumbar puncture, and echography are useful adjuncts in the diagnosis and management of VKH syndrome. Patients with this syndrome are treated generally with high dose systemic corticosteroids, immunomodulatory agents such as cyclosporine, or more recently biological response modifiers which are used as steroid-sparing agents to minizeminimize side effects of long term steroid use.

Since their discovery in the 1990s, biologic drugs have been used to treat uveitis refractory to traditional immunosuppressants. Many questions on their use though have remained unanswered; particularly when to initiate therapy, which agent and at what dosage to use, and for how long the treatment should continue.

The Biologic Response Modifiers represent the future of therapy in immune-mediated uveitis. Biological anti-inflammatory agents (for example antagonists of tumor necrosis factor alpha-like Infliximab and adalimumab) are also showing very promising results.

Biologics alone or combined with conventional therapies are used in refractory cases of Uveitis. Biologics reported for use in uveitis interferon alpha 2a (IFN-α 2a); anti-tumor necrosis factor (TNF) agents-infliximab and adalimumab; anti-interleukins (IL)-tocilizumab, secukinumab (in most of the published papers, this biologic has failed to demonstrate the ability to control uveitis when compared to placebo) and gevokizumab; anti-CD20-rituximab and anti-CD 25-daclizumab.

In many cases, these agents will be seen listed as the first choice in some autoimmune diseases, depending on the patient's history, age, sex, type and severity of the inflammatory disease, etc. The interdisciplinary treatment between ophthalmologists and rheumatologist is essential to initiate and monitor these therapies. Follow-up visits of subjects with uveitis should be aimed to determine the evolution of inflammatory signs until their complete resolution, thus ensuring the least possible consequences.

The most common side effects are localized site reactions (pain, erythema, and rash). other side effects include upper respiratory tract infections, urinary tract infections, cough, rash, back pain, nausea, vomiting, abdominal pain, headache, weakness, and fever. Other noted side effects include low or high blood pressure, chest pain, difficulty breathing, rash, itching, fever, and chills.

ELIGIBILITY:
Inclusion Criteria:

1. Uveitis with clinical features of Vogt-Koyanaga-Harada Syndrome.
2. A follow-up and assessment at least twelve months from the start of treatment.

Exclusion Criteria:

* Exclusion of other infectious and non-infectious uveiticuveitis etiologies that may mimic the given clinical presentation of autoimmune uveitis;
* The presence of contraindication to treatment with biologic drugs e.g. active or latent tuberculosis, viral hepatitis and demyelinating diseases.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Uveitis with clinical features of Vogt-Koyanaga-Harada Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
non-resolution of inflammation, or failure of complete clinical resolution of the primary lesion in cases of retinitis or choroiditis. | at 6 month
  Prospective
Recurrence of inflammation described as a two-step increase in inflammation as defined by the SUN working group criteria for anterior and intermediate uveitis | at 6 month
  prospective

SECONDARY OUTCOMES:
non-resolution of inflammation, or failure of complete clinical resolution of the primary lesion in cases of retinitis or choroiditis. | at 12 month
  prospective
Recurrence of inflammation described as a two-step increase in inflammation as defined by the SUN working group criteria for anterior and intermediate uveitis | at 12 month
  prospective

CONTACTS AND LOCATIONS:
Overall Officials: Salma Safwat, Master, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pasadhika S, Rosenbaum JT. Update on the use of systemic biologic agents in the treatment of noninfectious uveitis. Biologics. 2014 Feb 15;8:67-81. doi: 10.2147/BTT.S41477. eCollection 2014. PMID 24600203
- [Background] Fang W, Yang P. Vogt-koyanagi-harada syndrome. Curr Eye Res. 2008 Jul;33(7):517-23. doi: 10.1080/02713680802233968. PMID 18600484
- [Background] Rubsamen PE, Gass JD. Vogt-Koyanagi-Harada syndrome. Clinical course, therapy, and long-term visual outcome. Arch Ophthalmol. 1991 May;109(5):682-7. doi: 10.1001/archopht.1991.01080050096037. PMID 2025171
- [Background] Imrie FR, Dick AD. Biologics in the treatment of uveitis. Curr Opin Ophthalmol. 2007 Nov;18(6):481-6. doi: 10.1097/ICU.0b013e3282f03d42. PMID 18163000
- [Background] Hatemi G, Christensen R, Bang D, Bodaghi B, Celik AF, Fortune F, Gaudric J, Gul A, Kotter I, Leccese P, Mahr A, Moots R, Ozguler Y, Richter J, Saadoun D, Salvarani C, Scuderi F, Sfikakis PP, Siva A, Stanford M, Tugal-Tutkun I, West R, Yurdakul S, Olivieri I, Yazici H. 2018 update of the EULAR recommendations for the management of Behcet's syndrome. Ann Rheum Dis. 2018 Jun;77(6):808-818. doi: 10.1136/annrheumdis-2018-213225. Epub 2018 Apr 6. PMID 29625968